CLINICAL TRIAL: NCT02103413
Title: Multicenter Study of EUS-guided Biliary Drainage Versus Percutanenous Transhepatic Biliary Darinage for Malignant Biliary Obstruction After Failed ERCP
Brief Title: EUS-guided Biliary Drainage Versus Percutanenous Transhepatic Biliary Darinage for Malignant Biliary Obstruction After Failed ERCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Do Hyun Park, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EUS-BD-002
Record Dates: First submitted 2014-04-01; First posted 2014-04-03 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Cholestasis, Extrahepatic
MeSH Terms: conditions — Cholestasis, Extrahepatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS-BD (Experimental): EUS-BD using a fully or partially covered self-expanding metallic stent will be performed by EUS guided 19 G needle puncture.
  Interventions: Device: EUS-BD
- PTBD (Experimental): PTBD with 8.5F catheter will be inserted under fluoroscopic and/or ultrasonography guidance by experienced interventional radiologists.
  Interventions: Device: PTBD

INTERVENTIONS:
Device: EUS-BD — When the ERCP was unsuccessful, we tried one-step EUS-BDS using a linear-array echoendoscope (GF-UCT 240-AL 10 or AL 5, Olympus Medical Systems, Tokyo, Japan) at the same ERCP unit on the same session. EUS-BDS was performed by EUS-guided choledocoduodeostomy (EUS-CD) or EUS-guided hepaticogastrostomy (EUS-HG) at the discretion of involved endosonographers. Based on our modified protocol from two our proposed protocols, EUS-BD with transmural stenting was only considered.
  Arms: EUS-BD
Device: PTBD — PTBD was performed in selected patients with an 8.5F catheter inserted under fluoroscopic or ultrasound guidance by experienced interventional radiologists or endoscopists.
  Arms: PTBD

SUMMARY:
Although ERCP is almost always successful in patients with malignant biliary obstruction, selective biliary cannulation fails in some cases and conventional ERCP may not be possible in patients with tumor invasion of the duodenum or major papilla, surgically altered anatomy (e.g., Roux-en-Y anastomosis), or complex hilar biliary strictures. In such cases, percutaneous transhepatic biliary drainage (PTBD) is an useful alternative. However, PTBD had various complications and the presence of an external drainage catheter would also have a cosmetic problem related to the external drainage and an adverse impact on quality of life (QOL) of terminally ill patients.

Since endoscopic ultrasound-guided bile duct puncture was described in 1996, sporadic case reports of EUS-guided biliary drainage (EUS-BD) suggested that it was a feasible and effective alternative in patients with failed conventional ERCP stenting. The potential benefits of EUS-BD include one-stage procedure in ERCP unit, and internal drainage for avoiding long-term external drainage in cases where external PTBD drainage catheters cannot be internalized, thus significantly improving the QOL of terminally ill patients, and possibly lower morbidity than PTBD or surgery.

Up to date, only a few case series of EUS-BD with small numbers of patients have been published, and known the feasibility and safety in terms of the incidence of procedure-related clinical outcomes.10-21 There has been no comparative study between the outcomes of PTBD and EUS-BD focusing on the QOL, cost-effectiveness, and complications.

The researchers investigated the technical success of EUS-BD and PTBD in patients with malignant biliary obstruction after failed conventional ERCP as a prospective randomized comparative study in multicenters. Secondary endpoints were the cost-effectiveness and complications rates between EUS-BD and PTBD.

ELIGIBILITY:
Inclusion Criteria:

* Presence of unresectable malignant distal biliary obstruction (greater 2cm than distal to hilum, i.e., pancreatic cancer, common bile duct cancer, ampulla of Vater cancer, gallbladder cancer, duodenal cancer, and metastatic biliary obstruction)
* Failed conventional ERCP and inaccessible papilla because of accompanying duodenal obstruction, periampullary tumor infiltration, ampulla stenosis, or surgically altered anatomy (Billroth II operation, Roux-an-Y operation.)
* Histologic or cytologic diagnosis of malignancy, d) A Karnofsky index of ≧30%, e) No serious or uncontrolled medical illness
* Provided informed consent.

Exclusion Criteria:

* patient age of less than 18 years
* uncorrectable coagulopathy
* history of allergy to radiocontrast agents
* refusal to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Technical success of EUS-BD and PTBD | twelve months
  Technical success rate of EUS-BD and PTBD after failed ERCP

SECONDARY OUTCOMES:
Complications of EUS-BD and PTBD | twelve months
  Complications rate of EUS-BD and PTBD in patients who failed ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Do Hyun Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (2):
- South Korea (2):
  - Tae Hoon Lee, Cheonan
  - Woo Hyun Paik, Ilsan